CLINICAL TRIAL: NCT05528666
Title: Risk Perception in Multiple Sclerosis
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: COMB157G3001
Record Dates: First submitted 2022-09-02; First posted 2022-09-06 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Multiple Sclerosis
Keywords: Multiple sclerosis (MS),; Disease-modifying therapies (DMTs),; High efficacy treatments (HETs),; Nonhigh efficacy treatments (Non-HETs)
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (3):
- Overall cohort: Included all patients
- Previous Non-HET: Non-HETs include molecules classified as with moderate or modest efficacy such as: interferons, glatiramer acetate, dimethyl fumarate and teriflunomide.
  Interventions: Other: Non High Efficacy Therapy (Non-HET)
- Previous HET: HET include alemtuzumab, ofatumumab, ocrelizumab, natalizumab, cladribine, fingolimod and ozanimod.
  Interventions: Other: High Efficacy Therapy (HET)

INTERVENTIONS:
Other: High Efficacy Therapy (HET) — HET include alemtuzumab, ofatumumab, ocrelizumab, natalizumab, cladribine, fingolimod and ozanimod.
  Groups: Previous HET
Other: Non High Efficacy Therapy (Non-HET) — Non-HETs include molecules classified as with moderate or modest efficacy such as: interferons, glatiramer acetate, dimethyl fumarate and teriflunomide.
  Groups: Previous Non-HET

SUMMARY:
This study was a retrospective, non-interventional, cross-sectional, multi-cohort study of patients clinically diagnosed with RMS (RRMS and SPMS). Patients were classified according to the immediate previous treatment in two groups, those who were prescribed with high efficacy treatments (HETs) and those who were prescribed with non-high efficacy treatments (non-HETs). HET include alemtuzumab, ofatumumab, ocrelizumab, natalizumab, cladribine, fingolimod and ozanimod; and non-HETs include molecules classified as with moderate or modest efficacy such as: interferons, glatiramer acetate, dimethyl fumarate and teriflunomide.

DETAILED DESCRIPTION:
The study cohort consisted of RMS patients identified in the Adelphi Real World MS DSP, which was current up until the Q2/2021. The study was using waves VI-IX of the Adelphi DSP dataset.

Study period: Q1 2017 - Q1 & Q2 2021 (waves VI-IX of Adelphi DSP dataset).

Identification period: Q1 2017 - Q1 & Q2 2021 (waves VI-IX of Adelphi DSP dataset).

Index date: defined as the dates when the surveys were carried out (Q1 2017 - Q1 & Q2 2021).

ELIGIBILITY:
Inclusion Criteria:

* Patients included in the database with a diagnosis of RRMS and SPMS.
* Patients with current treatment at the index date.
* Patients with previous treatment at the index date.
* Patients to whom the physician decided to switch the treatment from the previous treatment to current treatment at the index date.
* Patients (males & females) with 18 years or older at index date.

Exclusion Criteria:

* Patients included in the database with the diagnosis of primary progressive MS (PPMS).
* Patients with other major neurological or psychiatric condition, which could potentially hinder the analysis.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study cohort consisted of RRMS and SPMS patients identified in the Adelphi Real World MS Disease Specific Program (DSP) (2017-2021) with a current and previous treatment at index date, and whose physician decided to switch their treatment.
Sampling Method: Non-Probability Sample
Enrollment: 4361 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2021-09-17 (Actual); Study Completion 2021-09-17 (Actual)

PRIMARY OUTCOMES:
Proportion of patients who were switched based on risk perception (infections, malignancies, others) | Throughout the study, approximately 5 years (2017 to 2021)
  Proportion of patients who were switched based on risk perception (infections, malignancies, others) were reported.

SECONDARY OUTCOMES:
Number of patients with ranking of the frequency of switches due to risk perception | Throughout the study, approximately 5 years (2017 to 2021)
  Proportion of patients who were switched based on risk perception (infections, malignancies, others) were reported.
Proportion of patients who switched due to lack of efficacy | Throughout the study, approximately 5 years (2017 to 2021)
  Proportion of patients who switched due to lack of efficacy due to new or enlarging lesions on MRI, increase in the frequency and/or severity of the relapses, progression in physical disability measured by EDSS or patient compliance issues between groups were reported.
Proportion of patients who changed treatment group versus patients who continued in the same treatment group | Throughout the study, approximately 5 years (2017 to 2021)
  Proportion of patients who changed treatment group versus patients who continued in the same treatment group were reported.
Number of relapses | Baseline
  Number of relapses were reported.
Expanded Disability Status Scale (EDSS) | Baseline
  The Expanded Disability Status Scale (EDSS) is a method of quantifying disability in multiple sclerosis and monitoring changes in the level of disability over time. The EDSS scale ranges from 0 to 10 in 0.5 unit increments that represent higher levels of disability.
Age | Baseline
  Age information reported
Gender | Baseline
  Gender information reported
Number of patients: Employment status | Baseline
  Patient employment status reported
Number of patients with Initial MS diagnosis | Baseline
  Number of patients with Initial MS diagnosis were reported.
Number of patients with Current MS diagnosis | Baseline
  Number of patients with Current MS diagnosis were reported.
Number of patients with previous disease modifying treatment | Baseline
  Number of patients with previous disease modifying treatment were reported.

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis Investigative Site, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Results for COMB157G3001 from the Novartis Clinical Trials Website — http://www.novctrd.com/ctrdweb/trialresult/trialresults/pdf?trialResultId=17971